CLINICAL TRIAL: NCT07402655
Title: A Study on the Epidemiology and Long-Term Functional Outcomes of Acute Traumatic Injuries to the Median, Ulnar, and Radial Nerves
Brief Title: Acute Traumatic Median, Ulnar, and Radial Nerve Injuries: Epidemiology and Long-Term Outcomes
Status: Recruiting | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Halenur Yaman, research assistant, Suleyman Demirel University
Other Study IDs: 104/15
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Nerve Damage; Trauma Nervous System
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ulnar nerve
  Interventions: Other: Peripheral Nerve Injury Assessment
- median nerve
  Interventions: Other: Peripheral Nerve Injury Assessment
- ulnar and median
  Interventions: Other: Peripheral Nerve Injury Assessment
- radial
  Interventions: Other: Peripheral Nerve Injury Assessment

INTERVENTIONS:
Other: Peripheral Nerve Injury Assessment — Standard clinical and functional assessment of acute traumatic peripheral nerve injuries, including motor, sensory, and functional outcome evaluations, without assignment to a specific therapeutic intervention.

SUMMARY:
Assessment of the Outcomes of Hand Nerve Injuries

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of acute traumatic peripheral nerve injury of the upper extremity (median, ulnar, radial, or combined injuries)
* Injury requiring surgical or conservative management
* Ability to provide informed consent

Exclusion Criteria:

* History of previous peripheral nerve injury or surgery in the affected upper extremity
* Presence of central nervous system disorders affecting upper extremity function
* Severe concomitant musculoskeletal injuries preventing functional assessment
* Inability to complete clinical and functional evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients presenting with acute traumatic peripheral nerve injuries of the upper extremity, including median, ulnar, radial, and combined nerve injuries, who are evaluated and managed at a tertiary care university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Michigan Hand Outcomes Questionnaire (MHQ) Total Score - Injured Hand | 6 months after injury
  Patient-reported hand outcomes assessed with the Michigan Hand Outcomes Questionnaire (MHQ) for the injured hand. Total score range: 0-100; higher scores indicate better hand-related outcomes.

SECONDARY OUTCOMES:
Grip Strength of Injured Hand (Jamar Dynamometer) | 6 months after injury
  Grip strength of the injured hand measured using a Jamar dynamometer (kg). Mean of 3 trials; higher values indicate greater strength.
Semmes-Weinstein Monofilament Test Threshold - Injured Hand | 6 months after injury
  Cutaneous pressure threshold assessed using Semmes-Weinstein monofilaments in the injured hand. Reported as monofilament level (or gram-force, if applicable); lower values indicate better sensation.
Static Two-Point Discrimination - Injured Hand | 6 months after injury
  Static two-point discrimination measured in millimeters (mm) in the injured hand; lower values indicate better discrimination.

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi Uygulama ve Araştırma Hastanesi, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No